CLINICAL TRIAL: NCT02917863
Title: Randomized Crossover Trial for the Evaluation of the Possible Effects in the Intestine of Two Different Pharmaceutical Forms of L - Thyroxine in Patients With Primary Acquired Hypothyroidism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Stefano Stagi, MD, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: THYR69; 2015-001248-12 (EudraCT Number)
Record Dates: First submitted 2016-09-07; First posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Microbiota; Thyroid hormone; L-Thyroxine; Celiac disease
MeSH Terms: conditions — Hypothyroidism; Celiac Disease | interventions — Thyroxine; Tablets; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solid L-Thyroxine (Experimental): Patients assume L-Thyroxine (tablet, per os) according to the Summary Product Characteristics for 6 months (then switch to the other formulation).
  Dosage in children with hypothyroidism:
  0-6 months: 10 mcg/kg body weight/die 6-12 months: 8 mcg/kg body weight/die
  1- 5 years: 6 mcg/kg body weight/die 5-10 years: 4 mcg/kg body weight/die
  Dosage in adults:
  initial dose of 50mcg/die; maintenance dose 100-200 (300) mcg/die (medium dose 2-2,5 mcg/kg body weight/die).
  Dosage will be adjusted according to TSH level.
  Interventions: Drug: L-Thyroxine (tablet, per os)
- Liquid L-Thyroxine (Active Comparator): Patients assume L-Thyroxine (oral drops, solution) according to the Summary Product Characteristics for 6 months (then switch to the other formulation).
  Dosage in children with acquired hypothyroidism:
  initial dose: 12,5-50 mcg/die maintenance dose: 100-150 mcg/m2 body surface area
  Dosage in adults:
  initial dose: 50 mcg/die; maintenance dose: 100-200 (300) mcg/die (medium dose 2-2,5 mcg/kg body weight/die).
  Dosage will be adjusted according to TSH level.
  Interventions: Drug: L-Thyroxine (oral drops, solution)

INTERVENTIONS:
Drug: L-Thyroxine (tablet, per os)
  Other Names: Eutirox
  Arms: Solid L-Thyroxine
Drug: L-Thyroxine (oral drops, solution)
  Other Names: Tirosint
  Arms: Liquid L-Thyroxine

SUMMARY:
Thyroid disorders, in particular hypothyroidism, are associated with gastrointestinal impairment, such as celiac disease. A study reported an increased prevalence of celiac disease in a large cohort of children affected by congenital hypothyroidism, underlying the relationship between these two conditions. The hypothesis of our study is that the onset of celiac disorder may be related to the gut concentration of thyroid hormone (TH) in hypothyroidism patients treated with replacement therapy. In fact, TH replacement therapy showed a low bioavailability with a consequent high gut concentration. Two different pharmaceutical formulations (liquid and solid, per os) are available. The liquid one has a better absorption profile and bioavailability than the solid; therefore, it is associated with a low TH intestinal concentration. According to our hypothesis, the solid TH formulation could increase the microbial diversity in the gut instead of the liquid form, due to the high local TH concentration. Based on these findings, the purpose of this study is to evaluate the effect of two different pharmaceutical formulations of TH on the gut in terms of modification of gut microbiota, inflammatory parameters and gut absorption.

ELIGIBILITY:
Inclusion Criteria:

* Children with primary acquired hypothyroidism that require Levothyroxine therapy (naïve patients, < 18 years)
* Informed consent from parents and patient

Exclusion Criteria:

* Age < 3 years
* Patients with secondary hypothyroidism, euthyroid sick syndrome or thyroid hormone resistant
* Patients with celiac disease, type I diabetes or other known autoimmune diseases
* Patients with genetic diseases or syndromes, such as Down, Williams-Beuren, Turner
* Assumption of antibiotics, probiotics, prebiotics, or other medications that could affect the gut microbiota in the month before the beginning of the study
* Gastrointestinal infectious diseases in the month before the beginning of the study
* Hypersensitivity to levothyroxine or any of the ingredients contained in the two pharmaceutical formulations
* Untreated adrenal insufficiency, untreated pituitary insufficiency and untreated thyrotoxicosis.
* Patients with cardiovascular disease
* Patients who show with impaired pancreatic function measured using the assay in faecal fat (steatocrit) at the screening visit

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Effects on gut inflammation parameter (Calprotectin) | 0-6-12 months
  Calculate the difference in gut inflammation parameter (calprotectin) among the two groups of patients at T6-T0 and T12-T6
Effects on gut absorption parameters | 0-6-12 months
  Calculate the difference in gut absorption parameters (Steatocrit) among the two groups of patients at T6-T0 and T12-T6
Effects on gut inflammation parameter (Osteoprotegerin) | 0-6-12 months
  Calculate the difference in gut inflammation parameter (osteoprotegerin) among the two groups of patients at T6-T0 and T12-T6
Effects on gut inflammation parameter (S100-A12 protein) | 0-6-12 months
  Calculate the difference in gut inflammation parameter (S100-A12 protein) among the two groups of patients at T6-T0 and T12-T6

SECONDARY OUTCOMES:
Baseline gut microbiota characterization | baseline
  Qualitative and quantitative (percentage) characterization of gut microbiota before the start of the therapy (T0)
Difference in gut microbiota among hypothyroid and healthy subjects | baseline
  Difference in gut microbiota among hypothyroid patients (T0) and healthy patients (data from Human Microbiome Project)
Incidence of deamidated AGA | 6-12-24 months
  Estimate the incidence of positive patients to deamidated AGA at T6, T12, T24 (follow-up)
Baseline gut inflammation parameters | baseline
  Evaluate gut inflammation (calprotectin, Osteoprotegerin and S100-A12 protein) parameters before the start of the therapy (T0)
Baseline gut absorption parameters | baseline
  Evaluate gut absorption (Steatocrit) parameters before the start of the therapy (T0)
Difference in Shannon Index in the gut microbiota among liquid and solid L-Thyroxine formulations | 0-6-12 moths
  Calculate the difference in Shannon Index (index of diversity) among the two groups of patients at T6-T0 and T12-T6
Difference in Chao I in gut microbiota among liquid and solid L-Thyroxine formulations | 0-6-12 moths
  Calculate the difference in Chao I (Species richness estimator) among the two groups of patients at T6-T0 and T12-T6
Difference in percentage of different species in gut microbiota among liquid and solid L-Thyroxine formulations | 0-6-12 moths
  Calculate the difference in percentage of different species (OTU, operational taxonomic unit) among the two groups of patients at T6-T0 and T12-T6

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stagi S, Manoni C, Cecchi C, Chiarelli F, de Martino M. Increased risk of coeliac disease in patients with congenital hypothyroidism. Horm Res Paediatr. 2011;76(3):186-92. doi: 10.1159/000328723. Epub 2011 Jul 15. PMID 21757873
- [Background] Smith DW, Klein AM, Henderson JR, Myrianthopoulos NC. Congenital hypothyroidism--signs and symptoms in the newborn period. J Pediatr. 1975 Dec;87(6 Pt 1):958-62. doi: 10.1016/s0022-3476(75)80918-8. PMID 1237554
- [Background] Robertson HM, Narayanaswamy AK, Pereira O, Copland SA, Herriot R, McKinlay AW, Bevan JS, Abraham P. Factors contributing to high levothyroxine doses in primary hypothyroidism: an interventional audit of a large community database. Thyroid. 2014 Dec;24(12):1765-71. doi: 10.1089/thy.2013.0661. PMID 25203248
- [Background] Sanchez E, Donat E, Ribes-Koninckx C, Fernandez-Murga ML, Sanz Y. Duodenal-mucosal bacteria associated with celiac disease in children. Appl Environ Microbiol. 2013 Sep;79(18):5472-9. doi: 10.1128/AEM.00869-13. Epub 2013 Jul 8. PMID 23835180
- [Background] Ianiro G, Mangiola F, Di Rienzo TA, Bibbo S, Franceschi F, Greco AV, Gasbarrini A. Levothyroxine absorption in health and disease, and new therapeutic perspectives. Eur Rev Med Pharmacol Sci. 2014;18(4):451-6. PMID 24610609
- [Background] Chao T, Wang JR, Hwang B. Congenital hypothyroidism and concomitant anomalies. J Pediatr Endocrinol Metab. 1997 Mar-Apr;10(2):217-21. doi: 10.1515/jpem.1997.10.2.217. PMID 9364356
- [Background] Guarner F, Malagelada JR. Gut flora in health and disease. Lancet. 2003 Feb 8;361(9356):512-9. doi: 10.1016/S0140-6736(03)12489-0. PMID 12583961